CLINICAL TRIAL: NCT03352492
Title: Effect of Peripheral Laser Iridotomy Placement on Post-operative Visual Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, Richard Trevino, OD, FAAO, Associate Professor, University of the Incarnate Word
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-02-003
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: Paired eye
Who Masked: Participant
Masking Description: Subject is masked to which eye has the iridotomy at which location
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral iridotomy: Superior (Experimental): Each subject in this single-arm study undergoes bilateral laser peripheral iridotomy surgery. Each participant will undergo superior laser peripheral iridotomy in one eye and temporal laser peripheral iridotomy in the fellow eye.
  Interventions: Procedure: Superior laser peripheral iridotomy
- Bilateral iridotomy: Temporal (Experimental): Each subject in this single-arm study undergoes bilateral laser peripheral iridotomy surgery. Each participant will undergo superior laser peripheral iridotomy in one eye and temporal laser peripheral iridotomy in the fellow eye.
  Interventions: Procedure: Temporal laser peripheral iridotomy

INTERVENTIONS:
Procedure: Superior laser peripheral iridotomy — Iridotomy placement between 11:00 and 1:00 o'clock
  Arms: Bilateral iridotomy: Superior
Procedure: Temporal laser peripheral iridotomy — Iridotomy placement at 3:00 or 9:00 o'clock
  Arms: Bilateral iridotomy: Temporal

SUMMARY:
To evaluate the influence of superior versus temporal laser peripheral iridotomy location on post-operative visual acuity and contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Angle-closure glaucoma
* Angle-closure glaucoma suspect

Exclusion Criteria:

* Monocular status
* Previous intraocular surgery
* Visual acuity worse than 20/40
* Prior episode of acute angle-closure glaucoma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity | 30 days post-operative
  Change from baseline best corrected visual acuity evaluated in number of letters correctly read on the ETDRS chart

SECONDARY OUTCOMES:
Change in Peli-Robson contrast sensitivity | 30 days post-operative
  Change from baseline in contrast sensitivity evaluated in number of letters correctly read on the Peli-Robson chart
Change in CSV-1000 contrast sensitivity | 30 days post-operative
  Change from baseline in contrast sensitivity evaluated using the number of correct responses on the CSV-1000 test

CONTACTS AND LOCATIONS:
Overall Officials: Richard Trevino, OD, Principal Investigator — University of the Incarnate Word
Locations (1):
- University of the Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No